CLINICAL TRIAL: NCT00314132
Title: Randomised, Double Blind, Multicentre, Placebo Controlled Phase III Study of the Safety and Tolerability Following Administration of Live Attenuated JE Vaccine (ChimeriVax™-JE)
Brief Title: Safety Study of ChimeriVax™-JE Vaccine to Prevent Japanese Encephalitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-040-010
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Encephalitis; Japanese Encephalitis
Keywords: Japanese Encephalitis; Encephalitis virus; ChimeriVax™-JE Vaccine
MeSH Terms: conditions — Encephalitis; Encephalitis, Japanese | interventions — Japanese Encephalitis Vaccines; ChimeriVax; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): All subjects received a single injection of placebo on Day 0.
  Interventions: Biological: 0.9% Saline
- ChimeriVax™ JE 4 log10 PFU Vaccine (Experimental): All participants received a single injection of ChimeriVax™ JE 4 log10 Plaque-forming unit (PFU) Vaccine on Day 0.
  Interventions: Biological: ChimeriVax-JE, Japanese Encephalitis vaccine

INTERVENTIONS:
Biological: ChimeriVax-JE, Japanese Encephalitis vaccine — 0.5 mL, Subcutaneous
  Other Names: ChimeriVax™
  Arms: ChimeriVax™ JE 4 log10 PFU Vaccine
Biological: 0.9% Saline — 0.5 mL, Subcutaneous
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess whether ChimeriVax™ JE vaccine (a new vaccine to be used for vaccination against Japanese encephalitis) is safe and well tolerated when compared to placebo (dummy) vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from the subject.
* Aged 18 years or above at screening.
* In good general health
* Subject available for the study duration
* For female subjects (of child bearing potential) a negative pregnancy tests at Screening and Day 0.

Exclusion Criteria:

* A history of vaccination against or infection with JE.
* Known or suspected immunodeficiency, use of immunosuppressive or antineoplastic drugs.
* History of thymoma, thymic surgery (removal) or myasthenia gravis.
* Clinically significant abnormalities on laboratory assessment
* Anaphylaxis or other serious adverse reactions characterised by urticaria or angioedema to foods, Hymenoptera (bee family) stings, or drugs including vaccines).
* Transfusion of blood or treatment with any blood product, including intramuscular or intravenous serum globulin within six months of the Screening Visit or up to Day 30.
* Administration of another vaccine or antiviral within 30 days preceding the Screening visit or up to Day 30.
* Physical examination indicating any clinically significant medical condition.
* Oral temperature >38°C (100.4°F) or acute illness within 3 days prior to inoculation.
* Intention to travel out of the area for an extended period that may affect the subjects ability to attend clinic visits prior to the study visit up to Day 30.
* Seropositive to hepatitis C virus (HCV) or HIV or positive for Hepatitis B Surface Antigen.
* Lactation or intended pregnancy in female subjects.
* Excessive alcohol consumption, drug abuse, significant psychiatric illness.
* A known or suspected physiological or structural condition that compromises the integrity of the blood-brain barrier (e.g. cerebrovascular disease, multiple sclerosis, trauma, infection, inflammation of the brain or meninges).
* Participation in another clinical study within 30 days of the screening visit for this study.
* Employee of the study site, Sponsor or Clinical Research Organization (CRO) involved with the management of the study.
* Any other reasons, which in the investigator's opinion, makes the subject unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2004 (Actual)
Dates: Start 2005-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Hull, MD, Principal Investigator — Vince and Associates Clinical Research
Locations (22):
- United States (16):
  - Burbank, California
  - Costa Mesa, California
  - Davis, California
  - San Francisco, California
  - Vallejo, California
  - Miami, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Bardstown, Kentucky
  - Livonia, Michigan
  - Sprnigfield, Missouri
  - Omaha, Nebraska
  - Winston-Salem, North Carolina
  - Fort Worth, Texas
- Australia (6):
  - Darlinghurst
  - Enoggera
  - Heidelbeg West
  - Kippa-Ring
  - Mill Park
  - Toorak Gardens

REFERENCES:
- [Derived] Torresi J, McCarthy K, Feroldi E, Meric C. Immunogenicity, safety and tolerability in adults of a new single-dose, live-attenuated vaccine against Japanese encephalitis: Randomised controlled phase 3 trials. Vaccine. 2010 Nov 23;28(50):7993-8000. doi: 10.1016/j.vaccine.2010.09.035. Epub 2010 Oct 8. PMID 20934459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and vaccinated from 10 October 2005 to 30 March 2006 at 6 clinical centers in Australia and 16 clinical centers in the US.
Pre-assignment Details: A total of 2004 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and vaccinated.
Groups:
- Placebo: Participants received a single injection of placebo on Day 0.
- ChimeriVax™-JE 4 log10 PFU Vaccine: Participants received a single injection of ChimeriVax™-JE 4 log10 Plaque-forming unit (PFU) Vaccine on Day 0.
Period: Overall Study
Arm/Group | Placebo | ChimeriVax™-JE 4 log10 PFU Vaccine
Started | 403 | 1601
Completed | 395 | 1583
Not Completed | 8 | 18
Not completed — Lost to Follow-up | 3 | 13
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ChimeriVax™-JE 4 log10 PFU Vaccine: Participants received a single injection of ChimeriVax™-JE 4 log10 PFU Vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | Placebo | ChimeriVax™-JE 4 log10 PFU Vaccine | Total
Number analyzed (Participants) | 403 | 1601 | 2004
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 403 | 1601 | 2004
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (14.12) | 34.6 (14.25) | 34.7 (14.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 721 | 886
  Male | 238 | 880 | 1118
Region of Enrollment [Number; unit: Participants]
  United States | 263 | 1201 | 1464
  Australia | 140 | 400 | 540

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment Related Adverse Events Post Vaccination With Either ChimeriVax™-JE or a Placebo
Description: Adverse events were collected by means of diary cards and scripted interviews. All adverse events reporting was considered "actively solicited" through Day 30.
Time Frame: Day 0 up to 30 days post-vaccination
Population: Treatment related adverse events were assessed in all participants who received an injection of study treatment, according to the treatment they received (Safety Population).
Measure: Number; unit: Participants
Groups:
- ChimeriVax™-JE 4 log10 PFU Vaccine: All participants received a single injection of ChimeriVax™-JE 4 log10 PFU Vaccine on Day 0.
Arm/Group | Placebo | ChimeriVax™-JE 4 log10 PFU Vaccine
Number analyzed (Participants) | 403 | 1601
Participants
  Fatigue | 90 | 365
  Malaise | 69 | 297
  Injection Site Pain | 36 | 199
  Feeling Hot | 27 | 152
  Chills | 17 | 112
  Injection Site Erythema | 14 | 74
  Injection Site Pruritus | 11 | 64
  Headache | 99 | 417
  Myalgia | 48 | 265
  Arthralgia | 21 | 119
  Diarrhea | 25 | 140
  Nausea | 26 | 114
  Abdominal Pain | 21 | 89
  Pharyngolaryngeal Pain | 10 | 55
  Dyspnea | 10 | 53
  Nasal Congestion | 9 | 14
  Nasopharyngitis | 13 | 10

2. Primary Outcome: Number of Participants Reporting Treatment Emergent Local Adverse Reactions and Treatment Emergent Systemic Reactions Post-vaccination With Either ChimeriVax™-JE or a Placebo
Description: Treatment emergent local adverse reactions: Injection Site Pain, Itching, Erythema, Swelling, Induration, Skin Rash, and others as reported.
  Treatment emergent systemic reactions: Malaise, Headache, Myalgia, Feeling Hot, Chills, Fatigue, Dyspnea, Wheezing, Nausea, Vomiting, Diarrhea, Abdominal Pain and others as reported.
Time Frame: Day 0 up to 30 days post-vaccination
Population: Treatment emergent local adverse reactions and systemic reactions were assessed in all participants who received an injection of study treatment, according to the treatment they received (Safety Population).
Measure: Number; unit: Participants
Arm/Group | Placebo | ChimeriVax™-JE 4 log10 PFU Vaccine
Number analyzed (Participants) | 403 | 1601
Participants
  Injection Site Pain | 36 | 199
  Injection Site Erythema | 15 | 74
  Injection Site Pruritus | 12 | 66
  Injection Site Hemorrhage | 4 | 21
  Injection Site Swelling | 4 | 17
  Injection Site Reaction | 3 | 10
  Injection Site Rash | 3 | 5
  Injection Site Induration | 0 | 1
  Injection Site Joint Pain | 0 | 1
  Injection Site Paresthesia | 1 | 0
  Injection Site Stinging | 0 | 1
  Injection Site Warmth | 0 | 1
  Fatigue | 112 | 479
  Malaise | 92 | 383
  Chills | 26 | 147
  Pyrexia | 7 | 26
  Headache | 124 | 597
  Myalgia | 67 | 352
  Arthralgia | 28 | 179
  Diarrhea | 36 | 183
  Nausea | 37 | 164
  Vomiting | 12 | 37
  Rash | 13 | 34

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from Day 0 to Month 6 post vaccination.
Arm/Group | Placebo | ChimeriVax™-JE 4 log10 PFU Vaccine
Serious Adverse Events (participants affected / at risk) | 2/403 | 5/1601
Other Adverse Events (participants affected / at risk) | 124/403 | 597/1601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=403) | ChimeriVax™-JE 4 log10 PFU Vaccine (N=1601)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Fallopian Tube Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=403) | ChimeriVax™-JE 4 log10 PFU Vaccine (N=1601)
Diarrhea (Gastrointestinal disorders) | 36 (42) | 183 (251)
Nausea (Gastrointestinal disorders) | 37 (50) | 164 (228)
Abdominal Pain (Gastrointestinal disorders) | 26 (33) | 138 (219)
Chills (General disorders) | 26 (38) | 147 (193)
Feeling Hot (General disorders) | 35 (55) | 193 (281)
Injection Site Pain (General disorders) | 36 (51) | 199 (279)
Malaise (General disorders) | 92 (150) | 383 (664)
Myalgia (Musculoskeletal and connective tissue disorders) | 67 (104) | 352 (561)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (44) | 179 (259)
Headache (Nervous system disorders) | 124 (251) | 597 (1253)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 23 (33) | 89 (122)
Fatigue (General disorders) | 90 (141) | 365 (699)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.